CLINICAL TRIAL: NCT07220993
Title: Novel Unedited Allo Cell Therapy For High Risk T-Cell Malignancies Using CD7-Specific Car Expressed On T Cells (NEO-CRIMSON)
Brief Title: Novel Unedited Allo Cell Therapy For High Risk T-Cell Malignancies Using CD7-Specific Car T Cells
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rayne Rouce, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-57819 - NEO CRIMSON
Record Dates: First submitted 2025-10-14; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: T-cell Acute Lymphoblastic Lymphoma; T-non-Hodgkin Lymphoma; T-cell Acute Lymphoblastic Leukemia
Keywords: Autologous CAR T cells; T-cell acute lymphoblastic lymphoma; T-non-Hodgkin lymphoma; T-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD7.CAR/28zeta T Cells (Experimental): Four dose levels will be evaluated. The T cells will be administered following lymphodepleting chemotherapy with cyclophosphamide and fludarabine.
  Interventions: Genetic: CD7.CAR/28zeta T Cells

INTERVENTIONS:
Genetic: CD7.CAR/28zeta T Cells — Fourdose levels will be evaluated:
  Dose level one: 1×10^7 cells/m^2 Dose level two: 3×10^7 cells/m^2 Dose level three: 5x10^7 cells/m^2 Dose level four: 1×10^8 cells/m^2

SUMMARY:
Patients eligible for this study have a type of blood cancer called T-cell leukemia or lymphoma (lymph gland cancer).

The body has different ways of fighting infection and disease. This study combines two different ways of fighting disease with antibodies and T cells. Antibodies are types of proteins that protect the body from bacterial and other diseases. T cells, or T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. Both antibodies and T cells have been used to treat cancer; they have shown promise, but have not been strong enough to cure most patients.

T cells can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study is called anti-CD7. This antibody sticks to T-cell leukemia or lymphoma cells because of a substance on the outside of these cells called CD7. CD7 antibodies have been used to treat people with T-cell leukemia and lymphoma. For this study, anti-CD7 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor.

In the laboratory, investigators have also found that T cells work better if they also add proteins that stimulate T cells, such as one called CD28. Adding the CD28 makes the cells grow better and last longer in the body, thus giving the cells a better chance of killing the leukemia or lymphoma cells.

In this study, investigators attach the CD7 chimeric receptor with CD28 added to it to T cells. Investigators will then test how long the cells last. These CD7 chimeric receptor T cells with CD28 are investigational products not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
Earlier, the patients previous bone marrow transplant donor gave the investigator blood to make CD7 CD28 chimeric receptor- T cells in the laboratory. These cells were grown and frozen for the patient. To get the CD7 antibody and CD28 to attach to the surface of the T cell, investigators will insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps investigators find the T cells in the patient's blood after investigators inject them. This virus also helps the investigators find the T cells in patients blood after they are injected. To ensure the T cells grow well in the lab, the investigators adds small amounts of medications that are often used to treat patients with cancer or other illnesses. These medications are washed off of the cells prior to injecting them into the patient's body. Because patients will have received cells with a new gene in them, patients will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. If patients cannot visit the clinic, they may be contacted by the research coordinator or physician.

When patients enroll on this study, they will be assigned a dose of CD7 chimeric receptor-T cells. Several studies suggest that the infused T cells need room to be able to proliferate (grow) and accomplish their functions and that this may not happen if there are too many other T cells in blood. Because of that, patients will receive two chemotherapy medications prior to receiving the CD7 chimeric receptor-T cells. One medication is called cyclophosphamide and the other fludarabine. Patients will receive 3 daily doses of each drug, ending at least one day before they receive the chimeric receptor-T cells. These drugs will decrease the numbers of the patients own T cells before investigators infuse the CD7 chimeric receptor T cells and also will help decrease the number of other cells that may interfere with the chimeric receptor-T cells working well. Although investigators do not expect any effect on tumors with the doses that patients will receive, these drugs are part of many regimens that are used to treat leukemia or lymphoma. Investigators prefer that patients do not receive other chemotherapy or treatments for their cancer until 6 weeks after cell infusion but patients can do so if their doctors thinks it is medically necessary.

Patients will be given an injection of cells into the vein through an IV at the assigned dose. Before patients receive the injection, they will be given a dose of Benadryl and Tylenol. The injection will take about 1-10 minutes. Investigators will follow patients in the clinic after the injection for up to 3 hours, and they will have to remain locally for at least 4 weeks after the infusion. If patients experience any side effects (see section on risks below), they may have to be hospitalized for evaluation and management. If after a 4-6 week evaluation period the patient has achieved a complete response (measured by bone marrow or radiology scans), the patient's primary oncology doctors may decide s/he should proceed to bone marrow transplant, at which time s/he will be removed from the treatment portion of the study.

The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

MEDICAL TESTS BEFORE TREATMENT

Before being treated, patients will receive a series of standard medical tests:

Physical exam and History Blood tests to measure blood cells, kidney and liver function Measurements of the patient's tumor by scans and/or bone marrow studies Testing of patient's blood for certain viral infections An ultrasound of patient's heart to make sure his/her heart function is appropriate for the study if the patient has not had one recently

MEDICAL TESTS DURING AND AFTER TREATMENT:

Patients will receive standard medical tests when they are getting the infusion and after:

Physical exams and History Blood tests to measure blood cells, kidney and liver function Measurements of the patient's tumor by scans and/or bone marrow studies 4-6 weeks after the infusion

To learn more about the way the CD7 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn. The total amount on any day is about 10 teaspoons (50 mL) or no more than 3 mL per 2.2 pounds body weight in children. This volume is considered safe but may be decreased if patients are anemic. This blood may be drawn from a central line if one is available. Blood will be taken before patients start the chemotherapy a few days prior to the cell infusion. On the day patients receive the cells, blood will be taken before the cells are given and several hours afterwards. Other blood will be drawn one week after the infusion, 2 weeks, 3 weeks, 4 weeks, 6 weeks and 8 weeks after the infusion, at 3 months, at 6 months, at 9 months, at 1 year, every 6 months for 4 years, then yearly for a total of 15 years. The total blood drawn during a patient's participation in this study will not exceed 280 teaspoons.

ELIGIBILITY:
Procurement Inclusion Criteria:

• Diagnosis of recurrent T-cell acute lymphoblastic leukemia (T-ALL), T-cell acute lymphoblastic lymphoma (T-LL), or T-non-Hodgkin Lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher))

AND

Relapsed post-allogeneic related donor (matched, mismatched, or haploidentical) HSCT from whom allogeneic CD7.CAR T cells can be manufactured.

AND

* suitable for allogeneic hematopoietic stem cell transplant (HSCT)
* with a suitable donor identified by a FACT accredited transplant center
* willing to proceed to transplant if the CD7.CAR treatment induces complete remission and the patient/donor remain suitable candidates.

Using NMDP donor assessment criteria, suitability is defined as "during the search process, a donor is fit to proceed to the next step- whether high-resolution or confirmatory HLA testing OR donor work-up." Documentation of suitability will be confirmed by the investigator prior to treatment.

*For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.

* CD7-positive tumor (≥20% CD7 positive blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory).
* Age ≤75 years old.
* Hgb ≥ 7.0 g/dL (can be transfused)
* Life expectancy greater than 12 weeks
* Patients must have an available partially-HLA matched allogeneic EBV-specific T cell line on a BCM IRB approved protocol which can be used as treatment in the event of uncontrolled EBV reactivation.
* Informed consent explained to, understood by and signed by patient/LAR. Patient/LAR given copy of informed consent.

Procurement Exclusion Criteria:

* Active infection requiring antibiotics
* Active infection with HIV
* History of other cancer (except non-melanoma skin cancer or in situ breast cancer or cervical cancer) unless the tumor was successfully treated with curative intent at least 2 years before trial entry.

Prior HSCT Donor Procurement Criteria:

• Donor must be prior hematopoietic stem cell transplant donor for patient relapsed post-allogeneic HSCT who meets patient screening eligibility criteria and has signed screening informed consent.

Prior transplant donors will be screened with the standard blood bank donor questionnaire, medical history, and testing for infectious disease markers (IDMs; which may be pending at the time of blood collection). Medical history may be obtained by the patient's primary/referring transplant team if collection is being done remotely. The physician assessment, donor questionnaire, and IDMs will be reviewed by the principal investigator or appropriate designee to confirm/provide final eligibility determination and documented in the donor's medical record.

• Informed consent explained to, understood by and signed by donor/LAR. Donor/LAR given copy of informed consent.

Treatment Inclusion Criteria:

• Diagnosis of recurrent T-cell acute lymphoblastic leukemia (T-ALL), T-cell acute lymphoblastic lymphoma (T-LL), or T-non-Hodgkin Lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher))

AND

Relapsed post-allogeneic related donor (matched, mismatched, or haploidentical) HSCT AND prior allogeneic donor available to donate blood for allogeneic CD7.CAR T-cell manufacture

AND

* suitable for allogeneic hematopoietic stem cell transplant (HSCT)
* with a suitable donor identified by a FACT accredited transplant center
* willing to proceed to transplant if the CD7.CAR treatment induces complete remission and the patient/donor remain suitable candidates.

Using NMDP donor assessment criteria, suitability is defined as "during the search process, a donor is fit to proceed to the next step- whether high-resolution or confirmatory HLA testing OR donor work-up." Documentation of suitability will be confirmed by the investigator prior to treatment.

*For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.

* CD7-positive tumor (≥20% CD7+ blasts or tumor cells by flow cytometry or immunohistochemistry (tissue) assessed in a CLIA certified Flow Cytometry/Pathology laboratory.
* Age ≤75 years old.
* Bilirubin less than 3 times the upper limit of normal.
* AST less than 5 times the upper limit of normal.
* Estimated GFR ≥ 50 mL/min.
* Pulse oximetry of > 90% on room air
* Karnofsky or Lansky score of ≥ 60%.
* Recovered from acute toxic effects of prior treatments (i.e. chemotherapy) at least one week before entering this study.
* ≥ 60 days post-allogeneic HSCT at time of treatment.
* Patients must have an available partially-HLA matched allogeneic EBV-specific T cell line on a BCM IRB approved protocol which can be used as treatment in the event of uncontrolled EBV reactivation.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
* Informed consent explained to, understood by, and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Exclusion Criteria:

* Currently receiving any investigational agents or having received any tumor vaccines within the previous 4 weeks.
* History of hypersensitivity reactions to murine protein-containing products.
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction (per investigator discretion).
* Clinically significant infection or uncontrolled viral reactivation of EBV, CMV, Adv, BK-virus, or HHV-6.
* Evidence of acute GVHD > Grade II or active chronic GVHD > mild global severity score.
* Currently taking corticosteroids for therapy at a dose of >0.5mg/kg prednisone equivalent.
* Patients who have received immunosuppressive treatment (IST) for GVHD within 28 days of infusion.
* Patients who have received donor lymphocyte infusion (DLI) within 28 days of infusion
* Any of the following cardiac criteria: Uncontrolled atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion; LVSF<30% or LVEF<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA III or IV. *Study requires cardiac echocardiography confirmation of absence of these conditions within 12 months of treatment.
* CNS abnormalities: Presence of CNS-3 disease defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm3 (unless negative by the Steinherz/Bleyer algorithm); Presence of any CNS disorder such as an uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage within the past 12 months, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate | 4 weeks
  Defined as the proportion of subjects in each group with DLT evaluated as per the CTCAE 5.0 with the exception of Cytokine Release Syndrome (CRS) and neurological toxicities that are related to T cell infusions.

SECONDARY OUTCOMES:
Overall Response Rate | 4 weeks
  Overall response rate is calculated as the proportion of subjects with the best overall response according to protocol defined response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rayne Rounce, MD, Principal Investigator — Baylor College of Medicine; LaQuisa Hill, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas